CLINICAL TRIAL: NCT02823353
Title: Fenofibrate in Combination With Ursodeoxycholic Acid in Primary Biliary Cirrhosis: a Randomized Control Study
Brief Title: Fenofibrate in Combination With Ursodeoxycholic Acid in Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Professor Consultant Physician, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20151230-4
Record Dates: First submitted 2016-01-28; First posted 2016-07-06 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2022-09

CONDITIONS: Primary Biliary Cirrhosis
Keywords: PBC; UDCA; Fenofibrate
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenofibrate + UDCA (Experimental): Fenofibrate (200 mg/day) in combination with ursodeoxycholic acid (13-15 mg/kg/day)
  Interventions: Drug: Fenofibrate; Drug: UDCA
- Monotherapy (Active Comparator): UDCA 13-15mg/kg/day
  Interventions: Drug: UDCA

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate 200mg/day
  Arms: Fenofibrate + UDCA
Drug: UDCA — UDCA 13-15mg/kg/day

SUMMARY:
Ursodeoxycholic acid (UDCA) has been the only treatment for primary biliary cirrhosis (PBC) approved by US and European drug administrations. Long-term use of UDCA(13-15 mg/kg/day) in patients with PBC improves serum liver biochemistries and survival free of liver transplantation However, about 40% of patients do not respond to UDCA optimally as assessed by known criteria for biochemical response. Those patients represent the group in need for additional therapies, having increased risk of disease progression and decreased survival free of liver transplantation. Both lab research and some clinical studies suggest that fenofibrate could improve cholestasis in multiple ways including reduce of bile acid synthesis, increase of biliary secretion and anti-inflammation effect. Here we start a random, open and parallel clinical research to explore the effect of fenofibrate in the PBC treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Patient with PBC defined by 2 in 3 of the following criteria: a.Positive antimitochondrial antibody type M2; b.Abnormal serum alkaline phosphatases (ALP > 1,5N) and aminotransferase (AST/ALT > 1N) activities; c.Histological hepatic injuries consistent with PBC.

Exclusion Criteria:

1. Pregnancy or desire of pregnancy.
2. Breast-feeding.
3. Co-existing liver diseases such as acute or chronic viral hepatitis, alcoholic liver disease, choledocholithiasis, autoimmune hepatitis, biopsy-proven non-alcoholic fatty liver disease, Wilson's disease and hemochromatosis
4. History or presence of hepatic decompensation (e.g., variceal bleeds, encephalopathy, or poorly controlled ascites).
5. History of urolithiasis, nephritis or renal failure (clearance of creatinine < 60 ml/mn).
6. Hepatotoxic drugs use before recruiting.
7. Fenofibrate anaphylaxis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Rate of patients with complete biochemical response | Week 48
  Normalization of alkaline phosphatase (ALP) or decrease of ALP by more than 40% compared to the baseline.

SECONDARY OUTCOMES:
Change in liver biopsy examinations according to conventional Ludwig system. | Week 48
  Histological evolution will be checked by liver biopsy at the end of the study to compare with baseline histological status. The Ludwig histological classification schemes will be used, which categorised the disease into four stages.
GLOBE risk scores at week 48. | Week 48
  The prognostic scores will be calculated at end of the study by GLOBE scoring system (proposed by Global PBC Study Group), which calculated based on serum values of bilirubin, ALP, albumin and platelet count after 1 year of UDCA therapy and age at baseline.
Change in liver stiffness status measured by magnetic resonance elastography. | Week 48
  The change of liver stiffness status at the end of the study compared to baseline checked by magnetic resonance elastography.
Change in serum levels of ALP compared to the baseline. | Weeks 0, 4, 8, 12, 24, and 48
  Absolute change in serum levels of ALP compared to the baseline.
Change in serum levels of bilirubin compared to the baseline. | Weeks 0, 4, 8, 12, 24, and 48
  Absolute change in serum levels of bilirubin compared to the baseline.
Change in serum levels of transaminase compared to the baseline. | Weeks 0, 4, 8, 12, 24, and 48
  Absolute change in serum levels of transaminase compared to the baseline.

OTHER OUTCOMES:
Change in pruritus. | Weeks 48
  The symptom of pruritus will be evaluated by questionnaire before enrolment and at the end of the study.
Change in fatigue. | Weeks 48
  The symptom of fatigue will be evaluated by Fatigue Impact Scale before enrolment and at the end of the study.
Change in serum Immunoglobulin M Levels. | Week 48
  Absolute change in serum levels of Immunoglobulin M compared to the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Liu Y, Guo G, Zheng L, Sun R, Wang X, Deng J, Jia G, Yang C, Cui L, Guo C, Shang Y, Han Y. Effectiveness of Fenofibrate in Treatment-Naive Patients With Primary Biliary Cholangitis: A Randomized Clinical Trial. Am J Gastroenterol. 2023 Nov 1;118(11):1973-1979. doi: 10.14309/ajg.0000000000002238. Epub 2023 Mar 9. PMID 36892506